CLINICAL TRIAL: NCT01422122
Title: The Effect of Vitamin D Supplementation on the Periodontal Health and Associated Outcomes in Pregnant Women
Brief Title: Study of Vitamin D Supplementation on Improvement of Gums Health
Acronym: VitaminD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Farhan Raza Khan, Consultant, Dentistry, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1479-Ped-ERC-10; Aga Khan University (Other: Aga Khan University, division of child and maternal health)
Record Dates: First submitted 2011-08-21; First posted 2011-08-23 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Gingival and Periodontal Disease; Deficiency of Vitamin D3; Pregnancy
Keywords: vitamin D; pregnancy; periodontal health; biomarkers
MeSH Terms: conditions — Periodontal Diseases | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): Oral vitamin D3 in syrup form
  Interventions: Drug: Vitamin D3
- placebo (Placebo Comparator): Placebo syrup identical in colour and taste to that of intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — 4000 mg per day, one tablespoon syrup per day
  Other Names: Vitamin D; Cholecaciferol
  Arms: Vitamin D
Drug: Placebo — one table spoon Syrup per day
  Other Names: placebo syrup
  Arms: placebo

SUMMARY:
There is a gap in knowledge regarding the effects of Vitamin D supplementation on periodontal status in pregnant wome. The investigators aim to evaluate the potential benefit, if any of vitamin D supplementation during pregnancy on periodontal disease and relevant outcomes including burden of infections and prematurity rates.

the investigators hypothesize that

1. Vitamin D supplementation during pregnancy improves the periodontal health.
2. There is an association between inflammatory biomarkers and periodontal health of pregnant females.
3. Vitamin D supplementation improves the outcomes of pregnancy such as prematurity rates and birth weight

DETAILED DESCRIPTION:
Periodontal disease is one of the most common chronic infectious diseases known to humans, with a reported prevalence varying between 10%-60% in adults. Periodontal health is commonly affected in pregnancy. The prevalence of pregnancy gingivitis varies widely, ranging from around 35%- 100%. Although, most of the periodontal changes during pregnancy are reversible but females with preexisting periodontitis or those who have metabolic disease such as diabetes may suffer increased periodontal destruction and may exhibit significantly greater probing pocket depth and attachment level. Periodontal disease, as a source of persistent infection, may induce systemic inflammatory responses that increase the risk of adverse pregnancy outcomes. However, so far the results have been mixed. As vitamin D metabolites may also alter the inflammatory response and have antimicrobial effects thus the use of vitamin D may affect periodontal status. Evidence is there which suggests that an association exists between low serum levels of Vitamin D and periodontal attachment loss. If the investigators take all of the above factors in consideration, the broad picture reveals that as vitamin D deficiency is prevalent in Pakistan, the pregnant females here are likely to have compromised periodontal health and probably poor pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females from 12-20 weeks of gestation who agree to participate in the study.
* Presence of at least 20 natural teeth in mouth excluding third molars.
* For controls: Non pregnant, healthy females matched with pregnant with respect to age and education.

Exclusion Criteria:

* Pregnant females with high Vitamin D levels,
* Women with metabolic diseases such as diabetes (type 1 or 2).
* Presence of acute dental or periodontal disease
* Presence of systemic disease and/or medication affecting the periodontium;
* Receipt of systemic antibiotic treatment or dental prophylaxis in the previous 3 months and those who do not provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Periodontal Probing Depth | 6 months
  Periodontal Probing Depth (PPD)is the distance between the gingival margin and the base of the pocket in millimeters). Clinical Attachment Loss (CAL) will also be determined (in mm)

SECONDARY OUTCOMES:
Interleukin 6 (IL-6) levels | 6 months
  Interleukin 6 (IL-6), is a biomarker of inflammation using CBA kit on Multiplex ELISA. Other biomarkers such as IL-2, IL-4, IL-10, TNF, IFN-ɣ and IL-17 will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, FRCPCH, PhD, Principal Investigator — Aga Khan University
Locations (1):
- AKU, Women & Child Health Outreach Office, Pind Dadan Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Khan FR, Iqbal NT, Ahmed K, Ahmad T, Hussain R, Bhutta ZA. Effect of Vitamin D Supplementation on the Salivary Cytokines of Pregnant Women: A Randomized Placebo-Controlled Trial. J Int Acad Periodontol. 2017 Oct 1;19(4):118-125. PMID 31473727